CLINICAL TRIAL: NCT00153985
Title: Multi-Center Study Using Allogeneic Stem Cell Transplantation Following Reduced Intensity Chemotherapy in Patients With Hemoglobinopathies
Brief Title: Allogeneic Stem Cell Transplantation Following Chemotherapy in Patients With Hemoglobinopathies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Massachusetts General Hospital (Other); Brigham and Women's Hospital (Other); Emory University (Other); Feist-Weiller Cancer Center at Louisiana State University Health Sciences (Other); Ohio State University (Other)
Responsible Party: Principal Investigator, Catherine Wu, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-338
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2013-03-12 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Hemoglobinopathies; Sickle Cell Disease; Thalassemia
Keywords: Hemoglobinopathies; Sickle cell anemia; sickle cell-hemoglobin C disease; sickle cell-B-thalassemia; transfusion-dependant thalassemia; allogeneic transplant; nonmyeloablative transplant; Stem cell transfusion; graft vs. host disease
MeSH Terms: conditions — Hemoglobinopathies; Anemia, Sickle Cell; Thalassemia; Hemoglobin SC Disease; Graft vs Host Disease | interventions — Busulfan; fludarabine; Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Busulfex — Given once daily for 4 days
Drug: Fludarabine — Given intravenously once daily for 4 days
Drug: Alemtuzumab — One day before fludarabine and busulfex are started, alemtuzumab will be given once daily for 5 days.
  Other Names: CAMPATH
Procedure: Stem Cell Transfusion — Performed three days after the end of chemotherapy

SUMMARY:
The purpose of this study is to determine if treatment with reduced-dose busulfex, fludarabine and alemtuzumab (CAMPATH) followed by sten cell infusion will allow for donor stem cells to grow in patients with hemoglobinopathies bone marrow and restore circulating blood counts. In addition the incidence and severity of side effects and of graft vs. host disease (GVHD) will be monitored.

DETAILED DESCRIPTION:
* In order to undergo transplant procedure, patients will be admitted to the hospital for approximately 10-14 days.
* To prepare patient's bone marrow to accept donor stem cells, they will receive fludarabine and busulfex. Fludarabine will be given intravenously once daily for 4 days. Busulfex will be given once daily for the same 4 days.
* One day before patients receive busulfex and fludarabine, they will also be given alemtuzumab intravenously once daily for 5 days.
* Three days after the end of chemotherapy, patients will receive the infusion of donor stem cells.
* If patients have thalassemia, they will receive subcutaneous injections of filgrastim starting on day one after the donor stem cell transfusion and will continue receiving filgrastim every day until it appears that the donor stem cells have been accepted. If the patient has sickle cell disease, filgrastim will not be given,
* Additional drugs will be given to help prevent infection (i.e. antibiotics).
* After stem cell infusion patients will be examined and have blood tests weekly for 1 month. Bone marrow biopsies, and blood work will also be performed 1 month, 3 months, 6 months and 1 year after stem cell infusion.
* Patients will be on the study for about 12 months. After study is completed progress will be monitored on an annual basis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sickle cell disease should have one or more of the following: acute chest syndrome requiring hospitalization; nonhemorrhagic stroke or central nervous system event lasting longer than 24 hours; recurrent caso-occlusive pain or recurrent priapism; sickle neuropathy; bilateral proliferative retinopathy and major visual impairment of at least one eye; osteonecrosis of multiple joints; transfusion dependence; vaso-occlusive.
* Patients with thalassemia should have one or more of the following: transfusion dependence; iron overload; presence of 2 or more alloantibodies against red cell antigens.

Exclusion Criteria:

* Pregnancy
* Acute hepatitis
* Cardiac ejection fraction < 30%
* Severe renal impairment
* Severe residual functional neurologic impairment
* Evidence of HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2004-03; Primary Completion 2008-03 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine J. Wu, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (6):
- United States (6):
  - Winship Cancer Institute-Emory University, Atlanta, Georgia
  - Feist-Weiller Cancer Center-LSU, Shreveport, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Ohio State University College of Medicine, Columbus, Ohio

REFERENCES:
- [Result] Armistead PM, Mohseni M, Gerwin R, Walsh EC, Iravani M, Chahardouli B, Rostami S, Zhang W, Neuberg D, Rioux J, Ghavamzadeh A, Ritz J, Antin JH, Wu CJ. Erythroid-lineage-specific engraftment in patients with severe hemoglobinopathy following allogeneic hematopoietic stem cell transplantation. Exp Hematol. 2008 Sep;36(9):1205-15. doi: 10.1016/j.exphem.2008.04.004. Epub 2008 Jun 11. PMID 18550258

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Activated for enrollment 3/4/2004. Closed to enrollment 4/25/2008. Participating institutions included: Dana-Farber Cancer Institute, Boston, Massachusetts, Feist-Weiller Cancer Center, LSU Health Sciences Center, Shreveport, Louisiana and Winship Cancer Institute, Emory University, Atlanta, Georgia
Pre-assignment Details: All enrolled patients received a stem cell transplant.
Groups:
- Transplant for Severe Hemoglobinopathies: Patients with severe hemoglobinopathies (eg. sickle cell disease, thalassemia major) with related donors who are identical at 6 HLA loci: (HLA-A, HLA-B, HLA-DRB1). The preparative regimen consisted of Busulfex, fludarabine and alemtuzumab.
Period: Overall Study
Arm/Group | Transplant for Severe Hemoglobinopathies
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Transplant for Severe Hemoglobinopathies
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 25 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Stable Engraftment With Donor Stem Cells in Patients With Severe Hemoglobinopathy.
Description: Outcome was measured by ANC >500 for three consecutive days prior to day 30 after PBSC infusion, >25% of hematopoietic cells are donor derived as determined by molecular chimerism assays or cytogenetic methods prior to day 45 after PBSC infusion and >25% of hematopoietic cells are donor derived as determined by molecular chimerism assays or cytogenetic methods after day 180 after PBSC infusion.
Time Frame: 3 years
Population: All patients enrolled.
Measure: Number; unit: participants
Arm/Group | Transplant for Severe Hemoglobinopathies
Number analyzed (Participants) | 2
participants | 2

2. Secondary Outcome: Solid Organ Toxicity Related to the Conditioning Regimen.
Description: Outcome was measured by the assessment of organ toxicity related to Busulfex, fludarabine and alemtuzumab.
Time Frame: 3 years
Population: All patients enrolled.
Measure: Number; unit: participants
Arm/Group | Transplant for Severe Hemoglobinopathies
Number analyzed (Participants) | 2
participants | 2

3. Secondary Outcome: The Incidence of Grade II-IV Acute Graft vs. Host Disease.
Description: Outcome was measured by incidence and severity of acute and chronic GVHD following donor stem cell infusion.
Time Frame: 3 years
Population: All patients enrolled.
Measure: Number; unit: participants
Arm/Group | Transplant for Severe Hemoglobinopathies
Number analyzed (Participants) | 2
participants | 2

ADVERSE EVENTS:
Time Frame: Through study completion in 2009 (or patient death)
Arm/Group | Transplant for Severe Hemoglobinopathies
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transplant for Severe Hemoglobinopathies (N=2)
Graft versus host disease (Immune system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transplant for Severe Hemoglobinopathies (N=2)
Infection (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No